CLINICAL TRIAL: NCT02159235
Title: Heavy Metals (Cadmium, Lead, Mercury, Zinc), Angiogenesis Factors (Endostatin, Angiostatin, VEGF) and Osteopontin in Patients With Coronary Artery Disease
Brief Title: Heavy Metals, Angiogenesis Factors and Osteopontin in Coronary Artery Disease (CAD)
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Jeanette Strametz-Juranek, Internal Medicine II-Cardiology, Medical University of Vienna
Other Study IDs: EK2010/910
Record Dates: First submitted 2012-12-05; First posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease; Heavy Metal Toxicity
Keywords: cadmium; lead; mercury; zinc; endostatin; angiostatin; VEGF; CAD; osteopontin
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Heavy Metal Poisoning

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AIHD-patients (ICD-10 I21): Patients suffering from acute ischemic heart disease according to ICD-10 I21
- CIHD-patients (ICD-10 I25): patients suffering from chronic ischemic heart disease according to ICD-10 I25

SUMMARY:
The present study aims is to investigate:

1. whether patients suffering from acute resp. chronic ischemic heart disease show higher levels for cadmium (Cd), lead (Pb) and mercury (Hg) than local and international reference levels suggest;
2. the correlation between severity of coronary artery disease and angiogenic and angiostatic factors (endostatin-ES, angiostatin-AS, VEGF-vascular endothelial growth factor, osteopontin-OPN) The patient population consists of about 270 female and male patients suffering either acute or chronic ischemic heart disease (AIHD:ICD-10 I21; CIHD: ICD-10 I25).
3. whether patients suffering CAD and valve calcification (mitral annulus, aortic valve) show higher levels of endostatin, angiostatin, osteopontin and VEGF compared to patients with CAD but without valve (annulus) calcification The measurement of cadmium (urine), lead, mercury, zinc, endostatin, angiostatin, VEGF (serum) and osteopontin (plasma) in patients with angiographically verified coronary artery disease are in the fore. Furthermore, basic laboratory diagnostics as well as data from coronary angiography and echocardiography will be collected. Additionally, the investigators will inquire heavy metal exposition during life by an interview.

Recruitment will be done during the in-patient stay at the General Hospital of Vienna, Medical University of Vienna.

DETAILED DESCRIPTION:
Patients with angiographically verified CAD of different severity were recruited at the Department of Cardiology, Medical University of Vienna. Detailed anamnestic and clinical data was collected incl. cardiovascular risk factor assessment, medication, ECG (electrocardiogram), routine laboratory parameters, echocardiography and all patients underwent an coronary angiography for diagnostic and/or therapeutic reasons on grounds of their underlying disease. The coronary artery system was divided into 17 segments and stenosis grade for each segment was measured. The segments were: left main, proximal/medial/distal LAD (lad left anterior descending artery), ramus circumflex, first and second marginal branch, posterolateral branch, first and second diagonal branch, proximal/medial/distal LCX (lcx left circumflex artery), proximal/medial/distal RCA (right coronary artery), ramus interventricular posterior and stenosis grade for each segment was measured. A simple 3-point-grading system ("Coronary Score") was developed considering both frequency and severity of CAD: 0 points for non-stenosed or only calcified segments, 1 point for each stenosis from <30-<50 %, 2 points for each stenosis from 50-<70 % and 3 points for each stenosis >70 %. Blood samples for determination of ES, AS and VEGF levels were taken at least two days before or after an acute event (angina pectoris, STEMI-ST-elevation myocardial infarction, NSTEM-Non ST-elevation myocardial infarction) or an invasive intervention (angiography). ES, AS and VEGF were analysed in serum, OPN in plasma by ELISA-Enzyme Linked Immunosorbent Assay according to the instructions of the manufacturer.

Echocardiography was performed to evaluate left and right ventricular function (multiple cross-sectional views), valve insufficiency/stenosis/calcification and wall movement disorders.

Hg and Pb levels were measured in full-blood, Cd in urine. The outcrop of full-blood samples for the determination of Pb and Hg was done by 2 ml ultrapure water and 2 ml nitric acid (68% sub-boiled). The sample aliquot was 0,5 ml, backfilling volume 20 ml. The determination of Pb and Cd was performed by ICPMS (inductively coupled plasma mass spectrometry) according to the ÖNORM EN ISO 17294-2. The determination of Hg was done by AFS (atomic fluorescence spectroscopy) according to the ÖNORM EN 17852. The outcrop of urine samples for the determination of Cd was done by 2 ml ultrapure water and 2 ml nitric acid (68% sub-boiled). The sample aliquot was 5 ml, backfilling volume 20 ml. The detection/quantification limits were 0,40/2 μg/l (Pb), 0,067/0,13 μg/l (Hg) and 0,12/0,40 μg/l (Cd). In case the quantification limit was undercut, the following expected amounts were used: Cd: 0,3 μg/l, Pb: 1 μg/l, Hg: 0,1 μg/l. In case of Cd and Hg Human-Biomonitoring (HBM)-I and II levels and in case of Pb reference levels from the German Environmental Agency.

Physical activity of the patients was defined/quantified as non physical activity, walking less 3h/week, walking more than 3 hours/week, sports less than 3 hours/week and sports more than 3 hours/week.

Statistical analysis was done with SPSS 20.0. Continuous and normally distributed data is described by means ± standard deviation (SD) and group differences are tested by independent sample t-test and correlation were calculated using Pearson's correlation coefficient. Continuous data with skew distribution or outliers is described ny median, first and third quartile and minimum and maximum. Group differences are tested by Mann-Whitney-U-test and correlations were calculated using Spearman's correlation coefficient. For data with values below the quantification limit a value below quantification limit was imputed (the same value for all these observations) and the non-parametric Mann-Whitney-U-test was used. All tests are performed two-sided and p-values ≤ 0,05 were considered significant. The protocol was approved by the Ethical Commission of the Medical University of Vienna and informed consent was obtained from patients.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering ICD-10 I21 or I25, age 18-80, female and male, non-smokers or ex-smokers for at least 7 years

Exclusion Criteria:

* no ICD-10 I21 or I25, patients younger that 18 or older than 80, smoking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be recruited during their in-patient stay at the General Hospital of Vienna
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
metal levels | 3 years
  Measurement of cadmium, lead, mercury and zinc in patients with acute or chronic ischemic heart disease (AIHD, CIHD).

SECONDARY OUTCOMES:
Correlation of endostatin-levels (ng/ml) with CAD-severity (Coronary artery score), valve calcification and grade of physical activity (as described in the methods) | 3 years
  Correlation of endostatin with severity of CAD (defined as described elsewhere) Correlation of endostatin with valve (annulus) calcification Correlation of endostatin with the grade of physical inactivity
Correlation of angiostatin levels (ng/ml) with CAD-severity (Coronary artery score), valve calcification and grade of physical activity (as described in the methods) | 3 years
  Correlation of angiostatin with severity of CAD (defined as described elsewhere) Correlation of angiostatin with valve (annulus) calcification Correlation of angiostatin with the grade of physical inactivity
Correlation of osteopontin-levels (ng/ml) with CAD-severity (Coronary artery score), valve calcification and grade of physical activity (as described in the methods) | 3 years
  Correlation of osteopontin with severity of CAD (defined as described elsewhere) Correlation of osteopontin with valve (annulus) calcification Correlation of osteopontin with the grade of physical inactivity
Correlation of VEGF-levels (ng/ml) with CAD-severity (Coronary artery score), valve calcification and grade of physical activity (as described in the methods) | 3 years
  Correlation of VEGF with severity of CAD (defined as described elsewhere) Correlation of VEGF with valve (annulus) calcification Correlation of VEGF with the grade of physical inactivity

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Strametz-Juranek, Univ.Prof.Dr, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria